CLINICAL TRIAL: NCT05353257
Title: A Randomized, Double-Blind, International Multicenter, Phase III Study to Evaluate the Anti-Tumor Efficacy and Safety of Serplulimab or Placebo in Combination With Chemotherapy and Concurrent Radiotherapy in Patients With Limited-Stage Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Serplulimab in Combination With Chemotherapy and Concurrent Radiotherapy in Patients With Limited-Stage Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-020-SCLC302
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Limited-Stage Small Cell Lung Cancer
Keywords: Limited-Stage Small Cell Lung Cancer; Serplulimab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; PE regimen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Serplulimab + carboplatin/cisplatin-etoposide + radiotherapy (Experimental): Participants will receive 4 cycles of standard-of-care chemotherapy (carboplatin/cisplatin-etoposide) plus Serplulimab 300 mg every 3 weeks (Q3W) concurrently with standard thoracic radiotherapy, with maximum 1 year after completion of cCRT or until disease progression, intolerable toxicity or other reasons specified in the protocol, whichever occurs first.
  Interventions: Drug: HLX10; Drug: carboplatin/cisplatin-etoposide; Radiation: Thoracic radiotherapy; Radiation: Prophylactic Cranial Irradiation (PCI)
- placebo + carboplatin/cisplatin-etoposide + radiotherapy (Placebo Comparator): Participants will receive 4 cycles of standard-of-care chemotherapy (carboplatin/cisplatin-etoposide) plus placebo every 3 weeks (Q3W) concurrently with standard thoracic radiotherapy, with maximum 1 year after completion of cCRT or until disease progression, intolerable toxicity or other reasons specified in the protocol, whichever occurs first.
  Interventions: Drug: carboplatin/cisplatin-etoposide; Radiation: Thoracic radiotherapy; Drug: Placebo; Radiation: Prophylactic Cranial Irradiation (PCI)

INTERVENTIONS:
Drug: HLX10 — Serplulimab is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  300mg Q3W
  Other Names: Serplulimab
  Arms: Serplulimab + carboplatin/cisplatin-etoposide + radiotherapy
Drug: carboplatin/cisplatin-etoposide — Etoposide: 100 mg/m2, IV, on Days 1, 2, and 3 of each cycle. Carboplatin: AUC = 5, IV, on Day 1 of each cycle up to a dose of 750 mg. investigator's choice.
  Cisplatin: 75mg/m2, IV, on Days 1 of each cycle. investigator's choice.
Radiation: Thoracic radiotherapy — Standard Thoracic Radiotherapy
Drug: Placebo — Placebo Q3W
  Arms: placebo + carboplatin/cisplatin-etoposide + radiotherapy
Radiation: Prophylactic Cranial Irradiation (PCI) — PCI will be strongly recommended for participants who achieve CR or PR after completion of chemoradiation treatment.

SUMMARY:
This study is a randomized, double-blind, multicenter, phase III clinical study to compare the clinical efficacy and safety of Serplulimab + chemotherapy+ concurrent radiotherapy vs chemotherapy+ concurrent radiotherapy in subjects with Limited-Stage Small Cell Lung Cancer.

DETAILED DESCRIPTION:
Eligible subjects in this study will be randomized to Arm A or Arm B at 1:1 ratio.

Arm A (Serplulimab arm): Serplulimab + chemotherapy(Carboplatin/Cisplatin-Etoposide)+concurrent radiotherapy; Arm B (placebo arm): Placebo + chemotherapy(Carboplatin/Cisplatin-Etoposide)+concurrent radiotherapy; The 4 stratification factors for randomization include: ECOG PS (0 or 1), staging (I/II or III), radiation fraction (bid or qd), and region (Asia or non-Asia).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years when signing the ICF.
2. Histologically diagnosed with SCLC.
3. Diagnosed with LS-SCLC (stage Ⅰ-Ⅲ of the AJCC 8th edition of the cancer staging), which can be safely treated with curative radiation doses.
4. Major organs are functioning well.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC.
2. Subjects suitable for surgery. Subjects who are suitable for surgery but refuse surgical treatment can be included.
3. Patients who have previously received systematic anti-tumor treatments for small cell lung cancer, including but not limited to radiotherapy, chemotherapy, and immunotherapy.
4. Patients with other active malignancies within 5 years or at the same time.
5. Subjects with known history of severe allergy to any monoclonal antibody.
6. Subjects with known anaphylaxis to carboplatin/cisplatin or etoposide.
7. In the judgment of the investigator, subjects who have any other factors that may lead to a premature discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to approximately 24months
  PFS, assessed by the Blinded Independent Central Review (BICR) as per RECIST v1.1
Overall survival (OS) | up to 36 months
  the time from randomization to death due to any cause

SECONDARY OUTCOMES:
Progression-free survival | up to approximately 24months
  PFS, assessed by the investigator as per RECIST v1.1
Objective response rate (ORR) | up to approximately 24months
  ORR, assessed by the BICR and investigator as per RECIST 1.1
Duration of remission (DOR) | up to approximately 24months
  DOR, assessed by the BICR and investigator as per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, MD, Principal Investigator — Shandong Cancer Hospital & Institute-department; Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (129):
- United States (31):
  - OPN-Glendale, Arcadia, California
  - OPN-Los Alamitos, Los Alamitos, California
  - Southern California Permanente Group, Los Angeles, California
  - Emad Ibrahim, MD, Inc, Redlands, California
  - Providence Medical Foundation, Santa Rosa, California
  - Lutheran Medical Center - Cancer Centers of Colorado, Golden, Colorado
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Advent Health Orlando, Orlando, Florida
  - Napa Research, Pompano Beach, Florida
  - Kansas University Mediacal Center, Fairway, Kansas
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Health Partners, Bloomington, Minnesota
  - Renown Health, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York City Health+HospitalsCorporation Elmhurst Hospital Center, Elmhurst, New York
  - Northwell Health, Queens, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Tricounty Hematology and Oncology Associates, Massillon, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Millennium Research & Clinical Development, Houston, Texas
  - Pro Research Tools, INC DBA Lumi Research, Kingwood, Texas
  - The University of Texas - Hope Cancer Center, Tyler, Texas
  - Innova Schar Cancer Insitute, Fairfax, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
- Austria (4):
  - Klinikum Klagenfurt am Worthersee, Klagenfurt
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Karl Landsteiner Institut für Lungenforschung und pneumologische Onkologie, c/o Klinik Floridsdorf Abteilung für Innere Medizin und Pneumologie, Vienna
  - Karl Landsteiner Institute for Lung Research and Pneumological Oncology, c/o Klinik Floridsdorf Department for Inner Medicine und Pneumology, Vienna
- China (63):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Gungzhouyikedaxuefushuzhongliuyiyuan, Guangzhou, Guangzhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hong Kong United Oncology Centre, Hong Kong, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - TaiHe Hospital Affiliated Hospital of Hubei University of Medicine, Shiyan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Zhongnan hospital of wuhan university, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First People's Hospital Of Changde City, Changde, Hunan
  - The Second Xiangya Hospita, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu people's Hospital, Yangzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Ganzhou Cancer Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shenyang The Tenth People's Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Tumor Hospital, Linyi, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Wenzhou University Hospital, Wenzhou, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second People's Hospital Of Yibin, Sichuan, Yibin
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Yuhang Branch of the First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The 1st Affiliated Hospital of WMU, Wenzhou, Zhejiang
- Czechia (10):
  - University Hospital Brno (Clinic For Lung Diseases and Tuberculosis), Brno
  - University Hospital Brno, Brno
  - University Hospital Olomouc (Oncology Clinic), Olomouc
  - University Hospital Ostrava (oncology department), Ostrava-Poruba
  - University Hospital Ostrava, Ostrava-Poruba
  - Nemocnice AGEL Ostrava-Vítkovice, Ostrava-Vitkovice
  - Nemocnice AGEL Ostrava-Vítkovice, Ostrava-Vítkovice
  - General University hospital in Prague (Oncology department), Prague
  - University Hospital Motol, Prague
  - University Hospital Motol (Pneumology Clinic 2.LF UK and FN Motol), Prague
- Germany (2):
  - Kliniken der Stadt Cologne GmbH, Cologne
  - University hospital Schleswig-Holstein, Travemünde
- Greece (2):
  - "Sotiria" Thoracic Diseases General Hospital of Athens, Athens
  - General Hospital of Athens "Alexandra", Athens
- Hungary (2):
  - Fejer County Szent Gyorgy University Teaching Hospital, Székesfehérvár
  - Pulmonary Institute of Torokbalint, Törökbálint
- Latvia (2):
  - Riga East University Hospital, Latvian Oncology Center, Riga
  - Clinic of Oncology, Pauls Stradins Clinical university hospital, Riga
- Netherlands (2):
  - Hospital St. Jansdal, Harderwijk
  - Isala Hospital, Zwolle
- Poland (2):
  - MedPoloniaSp. z o.o., Poznan
  - Lung and Chest Cancer Clinic, National Institute of Oncology, Warsaw
- Spain (9):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital German Trias i Pujol/ ICO Badalona, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Quironsalud Sagrado Corazón, Seville
  - Hospital Marques de Valdecilla, Valdecilla
  - University Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No